CLINICAL TRIAL: NCT06082960
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of GS-9911 as Monotherapy and in Combination With an Anti-PD-1 Monoclonal Antibody in Adults With Advanced Solid Tumors
Brief Title: Study of GS-9911 With or Without Antibody Treatment for Adults With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-521-6317
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: GS-9911 Monotherapy Dose Escalation (Experimental): Participants will receive escalating doses of GS-9911 monotherapy.
  Interventions: Drug: GS-9911
- Part B: GS-9911 Monotherapy Dose Expansion (Experimental): Participants will receive GS-9911 monotherapy at the recommended dose for expansion (RDE) determined in Part A.
  Interventions: Drug: GS-9911
- Part C: Dose Escalation: GS-9911 + Anti-PD-1 Monoclonal Antibody (Experimental): Participants will receive escalating doses of GS-9911 in combination with an anti-PD-1 monoclonal antibody (zimberelimab).
  Interventions: Drug: GS-9911; Drug: Zimberelimab
- Part D: Dose Expansion: GS-9911 + Anti-PD-1 Monoclonal Antibody (Experimental): Participants will receive GS-9911 at RDE determined in Part C in combination with an anti-PD-1 monoclonal antibody (zimberelimab).
  Interventions: Drug: GS-9911; Drug: Zimberelimab

INTERVENTIONS:
Drug: GS-9911 — Tablets administered orally
Drug: Zimberelimab — Administered intravenously
  Arms: Part C: Dose Escalation: GS-9911 + Anti-PD-1 Monoclonal Antibody; Part D: Dose Expansion: GS-9911 + Anti-PD-1 Monoclonal Antibody

SUMMARY:
The main goal of this first in human (FIH) study is to learn about the safety and dosing of GS-9911 when given alone or in combination with an anti-programmed cell death protein 1 (PD-1) monoclonal antibody in participants with advanced solid tumors.

The primary objectives of this study are to:

* Assess the safety and tolerability of GS-9911 as monotherapy and in combination with an anti-PD-1 monoclonal antibody in participants with advanced solid tumors
* Identify the maximum tolerated dose (MTD)/maximum administered dose (MAD) and the recommended dose for expansion (RDE) of GS-9911 as monotherapy and in combination with an anti-PD-1 monoclonal antibody in participants with advanced solid tumors

ELIGIBILITY:
Key Inclusion Criteria:

* Parts A, C, and D:

  * Participants with histologically or cytologically confirmed advanced solid tumors who have received, been intolerant to, or are ineligible for all treatments known to confer clinical benefit
* Part B:

  * Participants whose cancer previously derived clinical benefit from immune checkpoint inhibitors, or who have advanced solid tumor types for which immune checkpoint inhibitors are considered the standard of care and who have received, been intolerant to, or are ineligible for all treatments known to confer clinical benefit
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Evaluable (Part A) or measurable (Parts B, C, and D) disease as per Response Criteria Evaluation in Solid Tumors (RECIST) v1.1 criteria
* Adequate organ functions
* Tissue requirement:

  * Parts A-D: must be willing to provide baseline tumor tissue prior to enrollment
  * Part A backfill cohorts: a biopsy should be obtained prior to treatment and on treatment, if safely feasible
* Participants of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified methods of contraception

Exclusion Criteria:

* Positive serum pregnancy test or lactating female
* History of intolerance, hypersensitivity, or treatment discontinuation due to life- threatening immune-related adverse events on prior immunotherapy
* Receipt of the therapies listed below within the specified timeframe prior to planned Cycle 1 Day 1 including: major surgery (< 4 weeks), immunotherapy or biologic therapy (< 28 days), chemotherapy (< 21 days), targeted small molecule therapy (<14 days or 5 half-lives, whichever is sooner), hormonal or other adjunctive therapy (< 14 days), radiation therapy (< 21 days), live vaccine (< 28 days)
* Any prior allogeneic tissue/solid organ transplantation, including allogeneic stem cell transplantation
* Diagnosis of immunodeficiency, or requires systemic corticosteroids (> 10 mg of prednisone daily, or equivalent)
* History of autoimmune disease or active autoimmune disease that has required systemic treatment within 2 years prior to the start of study drug
* History of pneumonitis requiring treatment with corticosteroids, interstitial lung disease, drug-induced pneumonitis, or severe radiation pneumonitis (excluding localized radiation pneumonitis)
* Active second malignancy. Note: individuals with a history of malignancy that have been completed treated, with no evidence of active cancer for 2 years prior to enrollment, or individuals with surgically cured tumors with low risk of recurrence are allowed to enroll.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Symptomatic cardiovascular disease
* Active serious infection requiring ongoing treatment
* Active infection with hepatitis B virus (HBV), hepatitis C virus (HCV), or HIV.
* Symptomatic ascites or pleural effusion

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment-emergent Adverse Events | First dose date up to 90 days post last dose (up to 105 weeks)
Percentage of Participants With Treatment-emergent Serious Adverse Events | First dose date up to 90 days post last dose (up to 105 weeks)
Percentage of Participants Experiencing any Dose-limiting Toxicities (DLTs) in Dose-escalation Cohorts | First dose date up to 3 weeks

SECONDARY OUTCOMES:
Plasma Concentration of GS-9911 | Predose up to end of treatment (up to 105 weeks)
Pharmacokinetic (PK) Parameter: Cmax of GS-9911 | Predose up to end of treatment (up to 105 weeks)
  Cmax is defined the maximum observed plasma drug concentration.
PK Parameter: Tmax of GS-9911 | Predose up to end of treatment (up to 105 weeks)
  Tmax is defined as the time to maximum observed concentration.
Area Under the Concentration-Time Curve (AUC) of GS-9911 | Predose up to end of treatment (up to 105 weeks)
  AUC is defined as the area under the concentration versus time curve.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (4):
  - Smilow Cancer Hospital Phase 1 Unit, New Haven, Connecticut
  - SCRI Oncology Partners, Nashville, Tennessee
  - NEXT Oncology, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- University Health Network, Princess Margaret Cancer Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06082960